CLINICAL TRIAL: NCT01425034
Title: Postoperative Rehabilitation Following Trapeziectomy and Ligament Reconstruction Tendon Interposition: a Prospective, Randomized Multi-center Study
Brief Title: Postoperative Rehabilitation Following Trapeziectomy and Ligament Reconstruction Tendon Interposition
Acronym: LRTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Douglas Hutchinson, M.D., University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 49860
Record Dates: First submitted 2011-08-22; First posted 2011-08-29 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Osteoarthrosis of the Carpometacarpal Joint of the Thumb
Keywords: Cast; motion; thumb CMC arthritis; Collateral Ligament of Metacarpophalangeal Joint

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cast group (Active Comparator): The 'Cast' group will be placed in a thumb spica short arm cast with the thumb IP joint free. They will be allowed digit, thumb IP and elbow range of motion.
  Interventions: Other: casts for the thumb
- Motion group (Active Comparator): The 'Motion' group will be placed in a forearm based thumb spica splint with the thumb IP free. They will be allowed digit, thumb IP and elbow range of motion.
  Interventions: Other: Motion group

INTERVENTIONS:
Other: casts for the thumb — The 'Cast' group will be placed in a thumb spica short arm cast with the thumb IP joint free. They will be allowed digit, thumb IP and elbow range of motion.
  Other Names: Cast group
  Arms: Cast group
Other: Motion group — The 'Motion' group will be placed in a forearm based thumb spica splint with the thumb IP free. They will be allowed digit, thumb IP and elbow range of motion.
  Arms: Motion group

SUMMARY:
Carpometacarpal (CMC) arthritis of the thumb joint ('basal arthritis') is a common entity treated by hand surgeons in our society. It can be a significant source of functional disability secondary to a painful, and often weak, grip. Once patients have failed treatment by conservative means, such as splinting, anti-inflammatories, and cortisone injections, the next option is surgical management. Several surgical options are available depending on the severity of the disease. For the early stages of arthritis options include a ligament reconstruction or a metacarpal extension osteotomy. For advanced stages, only salvage procedures exist. These have included simple trapeziectomy, arthrodesis and implant arthroplasty. The most common procedure, however, has been a trapeziectomy with a ligament reconstruction tendon interposition

DETAILED DESCRIPTION:
Carpometacarpal (CMC) arthritis of the thumb joint ('basal arthritis') is a common entity treated by hand surgeons in our society. It can be a significant source of functional disability secondary to a painful, and often weak, grip. Once patients have failed treatment by conservative means, such as splinting, anti-inflammatories, and cortisone injections, the next option is surgical management. Several surgical options are available depending on the severity of the disease. For the early stages of arthritis options include a ligament reconstruction or a metacarpal extension osteotomy. For advanced stages, only salvage procedures exist. These have included simple trapeziectomy, arthrodesis and implant arthroplasty. The most common procedure, however, has been a trapeziectomy with a ligament reconstruction tendon interposition. During this procedure the arthritic trapezium is excised to remove arthritic joint surfaces, the anterior oblique ligament is reconstructed to restore thumb metacarpal stability and prevent axial shortening, and a fascial interposition is performed to reduce the likelihood of impingement between neighboring bones.

Postoperative rehabilitation and splinting protocols have varied widely between institutions. In fact, no studies have been published looking specifically at these protocols. Some institutions have taken a more conservative approach, having their patients immobilized by some means for up to twelve weeks with no motion for six weeks. Others advance their patients more quickly and start motion at four weeks with discontinuation of splinting at eight weeks.

There is one Cochrane Review on surgical treatment of trapeziometacarpal joint arthritis that compared seven surgical techniques. They looked at outcomes of pain, physical function, range of motion, global assessment, strength, CMC imaging and adverse effects. There was no mention of a therapy protocol.1

The Hand Clinics, a comprehensive, state-of-the-art review by experts in the field, provide current, practical information of the diagnosis and treatment of conditions affecting the hand and wrist. Each issue focuses on a single topic relevant to hand surgery practice. In the most recent arthritis issue, Clinics 26 (2010), Bodin et al. discussed many surgical techniques and alluded to therapy after eight weeks of casting but no specific protocol is defined. 2

A recent book publication by the American Society for Surgery of the Hand and the American Society of Hand Therapists include a chapter on arthritis incorporating rehabilitation interventions following soft tissue reconstruction of the CMC joint. They advocate a more conservative approach. Up to four weeks a forearm based thumb spica cast is utilized with thumb IP range of motion and edema control. At week 5 the patient is changed to a forearm based thumb spica splint with addition of active range of motion of the wrist and thumb MP and IP joints. CMC joint range of motion is started at week 6. At this point isometric strengthening to the wrist, thenar and first dorsal interosseous muscles is initiated. At week 10 patients begin light pinch and grip exercises. The splint is discontinued week 12.3

Hand therapists find the Diagnosis and Treatment Manual by the Hand Rehabilitation Center of Indiana to be the 'bible' of hand therapy. They advocate a more aggressive, earlier motion, protocol. At week 2, a forearm based thumb spica cast or splint is placed. At week 4 active and passive range of motion to the thumb and wrist is started including palmar and radial abduction, wrist flexion, extension, ulnar and radial deviation, and thumb circumduction, flexion, and extension. At week 6, gentle strengthening is begun with discontinuation of the splint.4

A less popular but frequently used book, Hand and Upper Extremity Rehabilitation, a practical guide, their chapter on Thumb CMC arthroplasty included a concise protocol similar to the Indiana protocol. At week 2, active and passive MCP and IP range of motion is started. At week 4, CMC abduction and extension, CMC opposition and wrist range of motion is started. At week 8, pinch and grip strength is stressed. There is no discussion about splinting. 5

Despite these published protocols, there have been no studies looking at which protocol is better. There have been no prospective, randomized trials comparing a conservative approach consisting of longer immobilization with a more aggressive approach advocating earlier motion and shorter splinting times.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 40 years old with basal arthritis who failed conservative treatment
* Patients receiving LRTI by one of three enrolled surgeons at the U or one of the two enrolled surgeons at Intermountain who consented to the study

Exclusion Criteria:

* Patients undergoing more procedures in addition to the LRTI that may alter the postoperative course, not including CTR or thumb MCP capsulodesis, MP fusion, trigger finger release
* h/o CRPS
* RA
* Revision LRTI

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2011-09; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
compare early motion vs. delayed motion after ligament reconstruction tendon interposition for thumb basal arthritis (LRTI) | 2 years
  DASH, VAS for pain, VAS for satisfaction, pinch and grip strength, coordination test and range of motion (thumb opposition)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Hutchinson, M.D,, Principal Investigator — University of Utah Orthopedics Center
Locations (1):
- InterMountain Health Care-TOSH orthopedic center, Murray, Utah, United States